CLINICAL TRIAL: NCT05689658
Title: Brazilian Diabetes Prevention Program: Pilot Study
Acronym: PROVEN-Dia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beneficência Portuguesa de São Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PROVEN-Dia
Record Dates: First submitted 2022-12-23; First posted 2023-01-19 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: PreDiabetes; Prediabetic State
MeSH Terms: conditions — Prediabetic State | interventions — Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brazilian Diabetes Prevention Program Group (Experimental): The program will be based on the American Diabetes Prevention Program (DPP), whose published results are used as a reference for prediabetic care patients in the Brazilian Diabetes Guideline. In order to reach the weight loss goal estimated at 0.5 to 1 Kg per week and 150 minutes of moderate physical activity per week, the program will offer individual and group visits, qualitative guidelines for improving diet, lifestyle and self-care.
  Interventions: Behavioral: Brazilian Diabetes Prevention Program
- Diet Group (Active Comparator): Diet prescription for weight loss
  Interventions: Behavioral: Diet

INTERVENTIONS:
Behavioral: Brazilian Diabetes Prevention Program — A Program structured in 7 visits (in group and individual) to guide the improvement of diet quality, self-care, and practice of physical activity
  Arms: Brazilian Diabetes Prevention Program Group
Behavioral: Diet — Hypocaloric diet prescription
  Arms: Diet Group

SUMMARY:
To structure a Brazilian Diabetes Prevention Program based on guidance for changing lifestyle promoted by the American Diabetes Prevention Program, using materials already developed by the Brazilian Ministry of Health and contextualizing it to the Brazilian Public Health System (SUS) and evaluating its effectiveness in a multicentric randomized clinical trial with 220 pre-diabetic patients and a follow up of 3 months. Outcomes are diet quality and time of physical activity. Health care professionals' perceptions regarding its incorporation into clinical practice will also be evaluated.

DETAILED DESCRIPTION:
This is a multicentric randomized clinical study coordinated by the Hospital Beneficência Portuguesa in São Paulo-Brazil and made possible by PROADI-SUS (SUS Institutional Development Support Program).

The study's objective is the Brazilian Diabetes Prevention Program development based on guidance for changing lifestyle promoted by the American Diabetes Prevention Program, using materials already developed by the Brazilian Ministry of Health and contextualizing it to the Brazilian Public Health System (SUS).

The program will not include a multidisciplinary orientation, but the prescription will have a multi-professional vision. The objective is to bring the multi-team together to discuss different aspects of the same intervention, such as accessibility, motivation, contexts, and needs, so that the program, to be guided by the nutritionist, can also be recognized and supported by the other teammates.

Once the program is defined, the research teams from the collaborating centers will be trained and qualified. 220 individuals with pre-diabetes will be included in the study and followed for 3 months. Outcomes are diet quality and time of physical activity. Health care professionals' perceptions regarding its incorporation into clinical practice will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index greater than or equal to 24kg/m2
* Have one of the following criteria: (CDC criteria for participating in the DPP)

  1. Diagnosis of prediabetes or
  2. Fasting blood glucose between 100-125mg/dl or blood glucose 2h after oral glucose tolerance test between 140 and 199mg/dl or HbA1c between 5.7 and 6.4% (maximum test date: last 3 months) or
  3. Previously diagnosed with gestational diabetes or
  4. High risk on the CDC prediabetes risk test
* With Internet access
* With personal cell phone access
* No prior nutritional monitoring (6 months)
* Live at least 60 minutes from the survey call center

Exclusion Criteria:

* Diagnosis of Diabetes Mellitus
* In secondary prevention for cardiovascular disease
* HIV patient with detectable viral load (amount of virus greater than 40 copies per ml of blood)
* Presence of illnesses that could seriously reduce your life expectancy or your ability to participate in the study
* Refuse to participate in the study (signing the Free and Informed Consent Form)
* Participation in another Randomized Clinical Trial whose objective interferes with the primary outcome of this research, such as diet quality and physical activity level
* Pregnant and lactating women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Quality of diet | 3 months
  to compare mean score of Brazilian Cardioprotective Nutritional Program dietary index (BALANCE DI) between groups. the index has a score from 0 to 40, with a high score indicating adherence to a healthy diet (BALANCE).
Minutes of Moderate Physical activity | 3 months
  to compare mean time in minutes of practice of moderate/vigorous physical activity over a week between groups

SECONDARY OUTCOMES:
Implementation Barriers and Facilitators | 3 months
  Identification of Barriers and Facilitators of Program implementation from a qualitative analysis approach. This is not a score on a scale. For the qualitative data, thematic content analysis will be performed with the transcription of the focus groups. This analysis will serve to describe and understand perceptions, interpretations and beliefs from the perspective of managers and professionals about the intervention. The thematic nuclei will be defined a posteriori according to the references of models and implementation frameworks also used for the realization of the focus groups
Moderate or vigorous physical activity (according to IPAQ-short) | 3 months
  to compare proportion of individuals who perform at the end of the follow-up moderate or vigorous physical activity
Cardioprotective diet adherence | 3 months
  to compare adherence to a healthy and cardioprotective diet based on the Cardiovascular Health Diet Index (CHDI) between groups. The CHDI had 11 components and a total score ranging from 0 to 110 points. the higher the score, the greater adherence to a healthy and cardioprotective diet
Global DNA Methylation | Baseline and 3 months
  participants' global DNA methylation using the RRBS method (Reduced Representation Bisulfite Sequencing).
weight | 3 months
  to compare mean weight (kg) between groups
HbA1c | 3 months
  to compare mean HbA1c(%) between groups
Glycemia | 3 months
  to compare mean Glycemia (mg/dL) between groups

CONTACTS AND LOCATIONS:
Locations (5):
- Brazil (5):
  - Hospital Universitário Professor Edgard Santos - HUPES, Salvador, Estado de Bahia
  - Hospital de Clínicas de Goiania, Goiânia, Goiás
  - Universidade Federal de Viçosa, Viçosa, Minas Gerais
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Universidade Federal do Tocantins, Palmas, Tocantins

IPD SHARING:
Plan to Share IPD: No